## Statistical Analysis Plan: SMART Project 3 (Efficacy Study)

Because these analyses will focus on determining and intervention feasibility and satisfaction, and preliminary intervention effect sizes (with less concern focused on testing for statistical significance), outcome analyses will be conducted using a separate analysis for each outcome at each follow up observation. To compare groups, baseline and follow up variables will be entered into a 5 (baseline vs. follow ups at 1, 2, 3, and 4 weeks) by 2 (CM vs. BSM) analysis of variance (ANOVA) which will yield effect sizes for time, and interactions of time by intervention. The primary dependent variables will be attendance at physician visits, saliva drug screen data (positive for buprenorphine and negative for illicit opioids), and prescription drug monitoring. We hypothesize that a greater number of CM participants will demonstrate adherence to buprenorphine-naloxone than BSM, but that those randomized to BSM will report increased time allocated to substance-free activities, decreased delayed reward discounting, and demand for opioid.